CLINICAL TRIAL: NCT06302504
Title: Nature-based Mindfulness Intervention Program for Family Caregivers with High Levels of Caring Related Stress
Brief Title: Nature-based Mindfulness Intervention Program for Family Carers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Hong Kong Polytechnic University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: Nature
Record Dates: First submitted 2024-03-04; First posted 2024-03-08 (Actual); Last update posted 2025-03-03 (Actual); Status verified 2025-02

CONDITIONS: Mental Health Issue
Keywords: caregiver; mindfulness-based program; nature

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Nature-based mindfulness program (Experimental): The program will include mindfulness exercises, including body scan, mindful stretching, mindful sitting, and befriending exercise. At least one of the four sessions will be conducted in retreat center in nature area.
  Interventions: Behavioral: Nature-based mindfulness program

INTERVENTIONS:
Behavioral: Nature-based mindfulness program — only one arm is included in this study

SUMMARY:
The program integrates ordinary mindfulness exercise with nature environment. Participants will be able to practice mindfulness in a natural environment in some of the program sessions. The study will study the effects of nature-based mindfulness program in reducing caregiving stress. The program will last for 4 session, 8 hours in total.

ELIGIBILITY:
Inclusion Criteria:

* parents with children experiencing divorce or separation
* parents of children with special needs
* family caregivers who are the primary caregivers of an older adult with dementia

Exclusion Criteria:

* parents or caregivers who cannot understand Cantonese version of Chinese
* parents or caregivers who have psychosis or developmental disabilities who are not able to comprehend the program

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 95 (Actual)
Dates: Start 2023-04-15 (Actual); Primary Completion 2024-03-31 (Actual); Study Completion 2024-05-31 (Actual)

PRIMARY OUTCOMES:
depression | Change from 1-month before intervention, pre-intervention, to 1-month follow-up, to 3-month after intervention
  measured by Depression Anxiety and Stress Scale (DASS-21)
anxiety | Change from 1-month before intervention, pre-intervention, to 1 month follow-up, to 3-month after intervention
  measured by Depression Anxiety and Stress Scale (DASS-21)
stress | Change from 1-month before intervention, pre-intervention, to 1-month follow-up, to 3-month after intervention
  measured by Depression Anxiety and Stress Scale (DASS-21)
family functioning | Change from 1-month before intervention, pre-intervention, to 1-month follow-up, to 3-month after intervention
  measured by The Family Adaptation, Partnership, Growth, Affection, Resolve Scale
family conflict | Change from 1-month before intervention, pre-intervention, to 1-month follow-up, to 3-month after intervention
  measured by The Conflict Tactics Scale
well-being | Change from 1-month before intervention, pre-intervention, to 1-month follow-up, to 3-month after intervention
  measured by The World Health Organization Well-being Index

CONTACTS AND LOCATIONS:
Locations (1):
- The Hong Kong Polytechnic University, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No
The funder decided not to share the data.